CLINICAL TRIAL: NCT00257933
Title: Oral Prednisolone Dosing in Children Hospitalized With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Joseph J. Zorc, M.D., The Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2005-9-4377
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2010-08-11 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Asthma
Keywords: Corticosteroids; Treatment; Pediatric
MeSH Terms: conditions — Asthma | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): High dose prednisolone
  Interventions: Drug: Prednisolone high dose
- 2 (Experimental): Lower dose prednisolone alternating with placebo
  Interventions: Drug: Prednisolone lower dose

INTERVENTIONS:
Drug: Prednisolone high dose — 4 mg/kg/day orally divided every 6 hours (maximum 30 mg per dose)
  Other Names: High Dose Prednisolone; Oral steriod; corticosteriods; asthma exacerbations
  Arms: 1
Drug: Prednisolone lower dose — 2 mg/kg/day orally divided q 12 (maximum 30mg/dose) alternating with placebo
  Other Names: Low dose Prednisolone; Oral prednisolone; Oral steriod; corticosteriods; asthma exacerbations
  Arms: 2

SUMMARY:
This study hopes to determine the appropriate oral steroid dose for treating children hospitalized with asthma exacerbations. Practice guidelines from different countries recommend a wide range of doses, and the doses used in actual practice vary widely. There is no data on what is the most appropriate dose of prednisone (or equivalent) in this situation. We will be looking at the dose recommended by the National Asthma Education and Prevention Program guidelines, which are published by the National Heart, Lung, and Blood Institute, as compared with a lower dose which is commonly used in practice. We hypothesize that the lower dose will be no worse than the higher dose as determined primarily by duration of hospitalization.

DETAILED DESCRIPTION:
Practice guidelines for the management of asthma in children universally recommend systemic corticosteroids for the treatment of moderate to severe asthma exacerbations. However, these guidelines vary widely with respect to dose, frequency, method of delivery, and duration of therapy. In actual practice, there is also considerable variation among clinicians in terms of corticosteroid dosing in children hospitalized with asthma exacerbations. At the Children's Hospital of Philadelphia (CHOP) the current standard is to use an initial dose of 4.0 mg/kg/day (1.0 mg/kg every 6 hours to a maximum of 30 mg/dose) although many other pediatric hospitals use a 2.0 mg/kg/day dose (1.0 mg/kg every 12 hours to a maximum of 30 mg/dose). Systematic reviews of the literature have called for a clinical trial to evaluate the effect of different doses of corticosteroids in treating pediatric asthma patients hospitalized with exacerbations.

This study will use a randomized, double-blind, controlled trial design in order to compare the efficacy of two different steroid doses in resolving acute exacerbations of asthma in hospitalized children. Children being hospitalized for asthma exacerbations from the CHOP emergency department (ED) will be eligible for study enrollment. Those that meet enrollment criteria will be randomized to receive prednisolone either in the higher dose (1.0 mg/kg (max 30 mg) every 6 hours), or the lower dose (1.0 mg/kg (max 30 mg) every 12 hours and placebo doses at 6 hour intervals in between) for the first 48 hours of hospitalization. Once 48 hours has past, all patients still hospitalized will receive 1.0 mg/kg (max 30 mg) every 12 hours for the duration of hospitalization. Approximately 156 patients with 78 in each arm of the study will be enrolled. This study should be completed in six to eight months. A non-inferiority study design will be used. The primary outcome will be duration of hospitalization, as determined by duration of time elapsed from first dose of prednisolone administered in the emergency department (ED) until the discharge dose of albuterol is administered. Secondary outcomes will include time elapsed from the time the admission order is written until the discharge order is written, time spent in each severity level of the asthma care pathway, degree and rate of improvement in forced expiratory volume in one second (FEV1), improvement in peak expiratory flows (PEF), improvement in asthma symptom scores, and rate of relapse after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma with at least two previous visits to ED or primary care provider for asthma care
* Clinical decision by ED attending physician to admit to Acute Care Unit (ACU) after standardized initial ED treatment

Exclusion Criteria:

* Clinical decision to begin continuous intravenous beta-agonist infusion
* Clinical decision to begin intravenous methylprednisolone therapy
* Clinical decision to admit to the Pediatric Intensive Care Unit
* Other concurrent disease such as sickle cell disease, cystic fibrosis, or cardiac disease
* Any contraindication to corticosteroid administration
* Any systemic corticosteroid treatment within two weeks of presenting to the ED
* Potential subjects will be excluded if informed consent is not obtained

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Zorc, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Prednisolone: High dose prednisolone: 1 mg/kg of oral prednisolone (maximum 30mg) every 6 hours
- Lower Dose Prednisolone: Lower dose prednisolone: 1 mg/kg (maximum 30mg)of oral prednisolone every 12 hours alternating with placebo
Period: Overall Study
Arm/Group | High Dose Prednisolone | Lower Dose Prednisolone
Started | 74 | 78
Completed | 74 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Prednisolone | Lower Dose Prednisolone | Total
Number analyzed (Participants) | 74 | 78 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 78 | 152
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.9 (4.4) | 7.0 (3.8) | 7.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 47 | 51 | 98
Region of Enrollment [Number; unit: participants]
  United States | 74 | 78 | 152

OUTCOME MEASURES:

1. Primary Outcome: Time Measured From the Administration of the Loading Dose of Prednisolone (2mg/kg up to Max 60mg) in the Emergency Department (ED) Until the Home Dose of Albuterol is Administered
Time Frame: Median time from loading dose to home dose of albuterol
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | High Dose Prednisolone | Lower Dose Prednisolone
Number analyzed (Participants) | 74 | 78
Hours | 35 [26 to 71] | 33 [25 to 51]

2. Secondary Outcome: Time Measured From the Writing of the Admission Order Until the Writing of the Discharge Order
Time Frame: Mean time from writing admit order until discharge order
Reporting Status: Not Posted
Measure: Number; unit: Hours

3. Secondary Outcome: Time Spent in Each Severity Level of the Asthma Care Pathway
Time Frame: Time spent in each severity level of pathway
Reporting Status: Not Posted

4. Secondary Outcome: The Rate and Degree of Change in Forced Expiratory Volume (FEV1) and Peak Expiratory Flow (PEF) Between Treatment Groups
Time Frame: Every 4 hours during hospitalization
Reporting Status: Not Posted

5. Secondary Outcome: Differences in Clinical Asthma Symptom Scores During Hospitalization Between Treatment Groups
Time Frame: Every 4 hours during hospitalization
Reporting Status: Not Posted

6. Secondary Outcome: Rate of Relapse Between Treatment Groups
Time Frame: 2 weeks after hospitalization
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Dose Prednisolone | Lower Dose Prednisolone
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/78
Other Adverse Events (participants affected / at risk) | 0/74 | 0/78

LIMITATIONS AND CAVEATS:
Limited ability to measure pulmonary function in hospitalized children with asthma did not allow measurement of this outcome.

Some protocol violations occurred

Single center study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No